CLINICAL TRIAL: NCT06903039
Title: NeoRes Study - Preoperative Chemotherapy in Colorectal Peritoneal Disease Prior to Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Acronym: NEORES
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEORES
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Metastatic; Peritoneal Metastases From Colorectal Cancer
Keywords: Colorectal cancer; Peritoneal metastases; Systemic chemotherapy; Chemotherapy sensitivity testing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Upfront Cytoreductive Surgery
- Neoadjuvant therapy First
- Conversion therapy first

SUMMARY:
Study Title:

Neores Study - Evaluating Systemic Chemotherapy Efficacy in Colorectal Peritoneal Metastases

Principal Investigator:

Peter Cashin Akademiska sjukhuset / Uppsala universitet

Background:

Peritoneal metastases from colorectal cancer are often associated with poorer outcomes compared to other metastatic sites. While systemic chemotherapy is widely used as a neoadjuvant treatment prior to CRS (Cytoreductive Surgery) and HIPEC (Hyperthermic Intraperitoneal Chemotherapy), its efficacy specifically for peritoneal metastases remains underexplored. Current practice in many countries includes neoadjuvant therapy to evaluate tumor biology and attempt tumor downstaging before surgery, despite the lack of robust data supporting this approach in colorectal cancer.

Purpose and Aims:

The study aims to evaluate how effective systemic chemotherapy is in treating isolated peritoneal metastases in colorectal cancer patients. The protocol defines two specific populations:

Patients receiving upfront systemic conversion chemotherapy. Patients undergoing open/close laparotomy (non-resectable disease found during surgery).

Key Research Questions:

What is the response rate to systemic chemotherapy before surgery? How many patients progress to CRS+HIPEC? What is the prognosis of those not undergoing surgery? How effective is FMCA (Fluorometric Microculture Cytotoxicity Assay) in predicting chemotherapy sensitivity? Do patients treated with FMCA-guided sensitive chemotherapy have better outcomes?

Methods:

This is a retrospective chart review study based on patient data from 2004-2021. It includes:

Review of HIPEC MDT (multidisciplinary team) conference notes to identify patients recommended for neoadjuvant conversion therapy.

Review of open/close laparotomy cases with FMCA testing.

Inclusion Criteria:

For HIPEC Pathway:

Colorectal cancer with isolated peritoneal metastases. Patients recommended for systemic chemotherapy before CRS+HIPEC.

For Open/Close Pathway:

Isolated peritoneal metastases discovered during surgery. Successful FMCA analysis performed.

Updated Inclusion (2024):

Patients with simultaneously resectable liver, para-aortal, and lung metastases are now allowed.

Exclusion Criteria (both pathways):

Appendiceal cancer. Retroperitoneal lymph node metastases. Other systemic metastases (liver, lung, brain, bone, etc.), unless resectable under updated criteria.

Data Collection:

Patient data will be retrieved from:

Uppsala University Hospital records Nationella Patientöversikten (national electronic health record) Swedish patient registry Swedish Colorectal Cancer Registry (SCRCR) (especially for molecular markers like KRAS, NRAS, BRAF, PIK3CA, MMR) When data is incomplete, referral hospitals will be contacted to gather additional information on administered chemotherapy (first and second-line therapies), therapy response, and survival outcomes.

Endpoints:

For chemotherapy group: Response to therapy and conversion to CRS+HIPEC. For open/close group: Progression-free survival and overall survival. Evaluation of FMCA sensitivity prediction accuracy. Outcomes based on whether patients received FMCA-indicated sensitive or resistant chemotherapy.

Statistical Methods:

Descriptive statistics. Kaplan-Meier survival curves. Cox proportional hazards models.

Clinical Significance:

There is a clear lack of high-quality evidence evaluating systemic chemotherapy's role in isolated peritoneal metastases. Despite being widely used, neoadjuvant therapy may not significantly improve survival outcomes in these cases, as seen in analogous ovarian cancer settings. The Neores study seeks to clarify the real-world effectiveness of this approach and to evaluate whether FMCA-guided treatment has clinical utility in predicting treatment success.

Given the uniqueness of Uppsala's long-standing use of FMCA, the study could provide important insights for patient selection and personalized therapy decisions.

DETAILED DESCRIPTION:
Neores Study: Evaluating Systemic chemotherapy efficacy in colorectal peritoneal metastases

Ansvarig forskare:

Peter Cashin Akademiska sjukhuset / Uppsala universitet

Research plan Background The effectiveness of systemic chemotherapy on peritoneal metastases is still rather poorly investigated. It is clear from randomized medical oncology trials that patients with peritoneal metastases from colorectal cancer do more poorly than other metastatic colorectal cancer. Currently, many countries use neoadjuvant therapy as a downstaging treatment or a test of tumor biology prior to selecting patients for CRS and HIPEC. However, very little is published concerning this treatment modality and its downstaging ability.

Purpose and aims The main aim of this research project is to evaluate the efficacy of systemic chemotherapy on isolated peritoneal metastases from colorectal cancer. Here are some specific aims.

Upfront systemic conversion chemotherapy:

1. What is the response rate of preoperative systemic conversion chemotherapy? 2. How many patients go on to CRS+HIPEC? 3. Those who do not come to surgery, what is their prognosis? Open/close laparotomy

1. How many patients have a successful FMCA test on chemotherapy sensitivity?
2. How many patients receive as first line chemotherapy a treatment that is sensitive vs resistant to given chemotherapy? Prognosis difference? Methods This will be a retrospective hospital charting study. The cohort will consist av two distinct populations - those that start with upfront systemic chemotherapy and those that come after an open/close laparotomy.

MDT pathway

1. Inclusion criteria HIPEC MDK where extensive isolated peritoneal metastases are noted Colorectal cancer Decision during HIPEC MDT to start systemic conversion chemotherapy
2. Exclusion criteria Appendiceal cancer Retroperitoneal lymph node metastases Other systemic metastases (e.g. liver, lung, brain, bone etc) Open-close surgery pathway

1. Inclusion criteria Colorectal cancer with isolated peritoneal metastases Going for upfront surgery, but resulting in an open/close laparotomy Successful FMCA analysis 2. Exclusion criteria Appendiceal cancer Retroperitoneal lymph node metastases Other systemic metastases (e.g. liver, lung, brain, bone etc) The first pathway will be evaluated by reviewing all HIPEC MDT conferences between 2004-2021. All patients with isolated peritoneal metastases from colorectal cancer that were sent for neoadjuvant conversion therapy will be identified. The clinical outcomes will be reviewed. The endpoints will be response to therapy and conversion rate to CRS+HIPEC.

The second pathway will be evaluated by reviewing all open/close patients with isolated peritoneal metastases from colorectal cancer. All patients with a successful FMCA analysis will be included for evaluation. The endpoint will be progression-free survival and overall survival.

Data will be taken from the Uppsala University Hospital charting as well as from the Swedish patient registry and from the "Nationella Patientöversikten" (a Swedish national digital charting service). If data on what chemotherapy was administered is not found through these sources, requests will be made to each respective referral hospital to send the oncology department charting in order to have complete data on what chemotherapy has been administered to each patient. Only the first and second-line therapies will be registered and the response to these therapies. Overall survival will also be registered.

Statistics Descriptive statistics, Kaplan-Meier curves and Cox proportional hazard modelling will be used to evaluate the respective endpoints.

Clinical significance Due to the paucity of published articles evaluating systemic chemotherapy in isolated peritoneal metastases, it is pertinent to investigate its use. Considering the fact that neoadjuvant treatment in the relatively chemotherapy sensitive ovarian cancer has not been proven to improve overall or recurrence-free survival, it seems logical that it may not have a relevant clinical use in the colorectal cancer situation. Despite this, neoadjuvant therapy is still widely used in colorectal cancer with peritoneal metastases. Furthermore, as the Uppsala institution has had the FMCA analysis available for chemotherapy sensitivity analyses for many years, this provides an opportunity to evaluate its predictive abilities for treatment outcome.

Publications Two papers are planned. The first paper will evaluate the neoadjuvant conversion chemotherapy use and the second paper will evaluate the FMCA analysis and its ability to predict response to systemic chemotherapy.

Updated research plan 2024 The aims have been added and updated in order to allow for immunotherapy evaluation.

1. Evaluate preoperative immunotherapy for colorectal cancer with peritoneal metastases (dMMR subtype)
2. Evaluate first-line palliative immunotherapy treatment of colorectal peritoneal metastases Inclusion criteria have been updated.

1: Simultaneous resectable liver, resectable para-aortal and resectable lung metastases are allowed.

Methods have been updated.

1: The project includes requisitioning data from the Swedish Colorectal Cancer Registry (SCRCR) in order to have more complete data on KRAS, NRAS, BRAF, PIK3CA, and MMR status. Also getting data on first-line treatment of colorectal cancer with peritoneal metastases is more complete from the SCRCR.

ELIGIBILITY:
Inclusion Criteria:

* HIPEC MDK where extensive isolated peritoneal metastases are noted
* Colorectal cancer
* Decision during HIPEC MDT to start systemic conversion chemotherapy

Exclusion Criteria:

* Appendiceal cancer
* Retroperitoneal lymph node metastases
* Other systemic metastases (e.g. liver, lung, brain, bone etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer with peritoneal metastases
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Overall survival | 24 months after treatment

SECONDARY OUTCOMES:
Objective response rate | 3 to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska Sjukhuset (Uppsala University hospital), Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be share upon reasonable request.